CLINICAL TRIAL: NCT04639674
Title: Prospective Randomized Study Evaluating the Efficacy of the Spherical Absorptive Carbon AST-120 in Hemodialysis Patients With Uremic Pruritus..
Brief Title: AST-120 in Hemodialysis Patients With Uremic Pruritus
Acronym: AST-120
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Conmed Pharmaceutical & Bio-Medical Corporation (Industry)
Collaborators: Tri-Service General Hospital (Other); Tungs' Taichung Metroharbour Hospital (Other); Chang Gung Memorial Hospital (Other); Taichung Veterans General Hospital (Other); Kaohsiung Medical University (Other); Taichung Tzu Chi Hospital (Other); Fu Jen Catholic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Conmed
Record Dates: First submitted 2020-10-27; First posted 2020-11-20 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Uremic Pruritus
MeSH Terms: interventions — AST 120

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AST-120 (Experimental): sachet Three times a day. (2g/pack*3pack/box)
  1 month
  Interventions: Drug: AST-120
- Control (No Intervention): No intervention

INTERVENTIONS:
Drug: AST-120 — If no other medicines are taken usually, take AST-120 one hour after each meal with a frequency of three doses a day and one dose every administration. The drug will be taken for four weeks.
  Other Names: Kremezin
  Arms: AST-120

SUMMARY:
The prevalence of cutaneous pruritus among hemodialysis patients is about 50% to 80%. There is only a handful of studies on the itchy skin of hemodialysis patients and the findings are to be validated. Effective drugs to treat cutaneous pruritus are not available yet. Hence, the purpose of the study is to eliminate the uremic toxins from the intestinal tract using AST-120 as a treatment measure to improve the symptom of the hemodialysis patients' cutaneous pruritus and discuss and assess its effectiveness. For this, the investigators will recruit 150 patients to validate the application potential of the AST-120 in the cutaneous pruritus brought about by uremia.

DETAILED DESCRIPTION:
Uremic toxins, such as indoxyl sulfate (IS) and p-cresol, or p-cresyl sulfate (PCS), are markedly accumulated in the organs of chronic kidney disease (CKD) patients. These toxins can induce inflammatory reactions and enhance oxidative stress, prompting glomerular sclerosis and interstitial fibrosis, to aggravate the decline of renal function. Consequently, uremic toxins play an important role in the worsening of renal and cardiovascular functions. Furthermore, they destroy the quantity and quality of bone. Oral sorbent AST-120 reduces serum levels of uremic toxins in CKD patients by adsorbing the precursors of IS and PCS generated by amino acid metabolism in the intestine. Accordingly, AST-120 decreases the serum IS levels and reduces the production of reactive oxygen species by endothelial cells, to impede the subsequent oxidative stress. This slows the progression of cardiovascular and renal diseases and improves bone metabolism in CKD patients. Although large-scale studies showed no obvious benefits from adding AST-120 to the standard therapy for CKD patients, subsequent sporadic studies may support its use.

Pruritus is a common and distressing symptom that affects patients with chronic kidney disease (CKD). Indoxyl sulfate (IS) and p-cresyl sulfate (PCS) are uremic toxins with similar protein binding, dialytic clearance, and proinflammatory features. The pathogenesis of uremic pruritus is not well elucidated, although it is theorized that inflammation may play a role. Elevated levels of C-reactive protein (CRP), interleukin-6, and interleukin-2 have been found among patients on hemodialysis suffering from pruritus, which may also partly explain the association the investigators found between low hemoglobin levels and a higher prevalence of pruritus, given the association between low hemoglobin and inflammatory states. Since the pathophysiology of uremic pruritus is multifactorial. Subclinical or overt uremic neuropathy, skin or nerve inflammation in the context of kidney failure-associated chronic systemic inflammation, or an increase in activity of μ-opioid receptors due to kidney failure have all been implicated.

A large, international study demonstrated the prevalence of moderate-to-extreme pruritus among patients with end-stage kidney disease on hemodialysis to be approximately 40% and was associated with a higher prevalence of comorbid conditions, worse biochemical profiles, poorer mental and physical quality of life, a higher probability of depression, and poorer sleep quality and survival. More recently, this prevalence was shown to range from 26% in Germany to 48% in the United Kingdom. Other studies have also demonstrated an association between pruritus and worse kidney disease burden scores, poorer health-related quality of life, and greater frequency of sleep disturbances in patients on dialysis.

However, pruritus is often overlooked by health care providers within dialysis units. In dialysis facilities where 21%-50% of patients reported having severe pruritus, only 1% of medical directors estimated this same prevalence. This may be due, in part, to underreporting by patients, as 17% of patients who were nearly always or always bothered by pruritus had not reported their symptoms to any health care provider.

Uremic pruritus intensity is also associated with multiple health-related quality-of-life outcomes, such as sleep quality, mood, and social function, and is independently associated with mortality. Uremic pruritus has been identified as a key research priority by patients with kidney disease.

Although several small studies have examined a variety of interventions, the efficacy of these interventions and the optimal treatments remain poorly defined. To address this important knowledge gap, the investigators systematically reviewed the literature and summarized the evidence for the major interventions for the treatment of uremic pruritus. The investigators will choose AST-120 as therapeutic agents for uremic pruritus.

ELIGIBILITY:
Inclusion Criteria:

1. Age of the subject: Over 20 (incl.) to less than 100
2. The patient must have undergone regular hemodialysis (excluding Hemodiafiltration or HDF) three times a week for at least six consecutive months and the Kt/V value, an indicator of the hemodialysis efficiency measured by urea nitrogen reduction ratio, must be greater than 1.2.
3. The patient must have taken drugs for the treatment of the cutaneous pruritus within the past six months and the effectiveness is not significant.
4. The patient must have not used AST-120 within the past three months.
5. The average VAS (Visual Analogue Scale) score of three itchy skin assessments during the screening period must be greater than or equal to 4 (VAS≧4).
6. Stable hemodialysis fistulas (both Arteriovenous Fistula, Arteriovenous Graft) must be available.
7. The patient must cooperate in the implementation of the investigational drug administration plan.
8. The patient must be able to sign the Informed consent form correctly.
9. The patient must be able to communicate with the researchers and understand the details of the study project.
10. All the drugs that the patient has taken must be traceable to a prescription.

Exclusion Criteria:

1. A physician has advised the patient not to take AST-120.
2. The patient suffers from poorly controlled high blood pressure, liver disease (higher than the liver function index ALanine aminoTransferase by 2.5 times or more), cholestasis, heart disease (congestive heart failure, coronary heart disease, ischemic heart disease), brain stroke, malignant tumor, acute inflammation, acute infection, or active lung disease.
3. The patient suffers from any skin disease not attributable to uremic toxins, including allergic or mycotic dermatitis. (If necessary, visit a dermatologist for diagnosis.)
4. The serum calcium level is higher than 10.5 mg/dl, serum phosphorus level is higher than 6.5 mg/dl, hemochrome level less than 9.0 g/dl, or serum parathyroid hormone level higher than 600 pg/ml.
5. The patient is pregnant or nurses a baby.
6. The formula of the drug for cutaneous pruritus has been changed 2 weeks before the screening.
7. The skin has undergone UV irradiation or acupuncture therapy 6 weeks before the screening.
8. Excessive alcohol or drug abuse has occurred 12 weeks before the screening.
9. The patient has participated in an interventional clinical trial 2 months before the screening.
10. The patient of the clinical trial may not accept any antibiotic treatment during the screening and trial period (because antibiotics will affect the concentration of the uremic toxins).
11. The patient suffers from digestive tract motility disorder and peptic ulcer disease or esophageal varices.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-07-02 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Visual analog scale | Change From Baseline in VAS at 2 Months
  Symptoms of skin itching: Visual analog scale (VAS)

SECONDARY OUTCOMES:
5-D itch scale | Change From Baseline in Scale at 2 Months
  Symptoms of skin itching: 5-D itch scale
Hospital Anxiety and Depression Scale | Change From Baseline in Scale at 2 Months
  Emotional stress: Hospital Anxiety and Depression Scale (HADS),
Center for Epidemiologic Studies Short Depression Scale | Change From Baseline in Scale at 2 Months
  Depression Scale (CES-D-R10)(Note, CES-D-R10 is conducted only at one center.)
Kidney Disease Quality of Life Scale | Change From Baseline in Scale at 2 Months
  Kidney Disease Quality of Life (Quality of Life Instrument / KDQOL) (Note, KDQOL is conducted only at one center.)
Urine toxin index | Change From Baseline in index at 2 Months
  Serum indoxyl sulfate (IS) / p-cresyl sulfate (PCS)
Aspartate transaminase (AST) | Change From Baseline in biochemical indicators at 2 Months
  Biochemical indicators
Creatinine | Change From Baseline in biochemical indicators at 2 Months
  Biochemical indicators
Urea nitrogen (BUN) | Change From Baseline in biochemical indicators at 2 Months
  Biochemical indicators
Blood calcium | Change From Baseline in biochemical indicators at 2 Months
  Biochemical indicators
Blood phosphorus | Change From Baseline in biochemical indicators at 2 Months
  Biochemical indicators
Albumin | Change From Baseline in biochemical indicators at 2 Months
  Biochemical indicators
Hemoglobin | Change From Baseline in biochemical indicators at 2 Months
  Biochemical indicators
White blood cell count | Change From Baseline in biochemical indicators at 2 Months
  Biochemical indicators
Parathyroid hormone | Change From Baseline in biochemical indicators at 2 Months
  Biochemical indicators
High-sensitivity C-reactive protein (hsCRP) | Change From Baseline in inflammation indicators at 2 Months
  Inflammation indicators
Interleukin-6 | Change From Baseline in inflammation indicators at 2 Months
  Inflammation indicators
Tumor necrosis factor-α | Change From Baseline in inflammation indicators at 2 Months
  Inflammation indicators
Beta2-microglobulin | Change From Baseline in inflammation indicators at 2 Months
  Inflammation indicators

CONTACTS AND LOCATIONS:
Overall Officials: Po-Sung Lin, Dr., Study Chair — Tungs' Taichung MeltroHarbor Hospital; Chia-Chao Wu, Dr., Study Chair — Tri-Service General Hospital; Shou-Hsuan Liu, Dr., Study Chair — Chang Gung Memorial Hospital; Yi-Wen Chiu, Dr., Study Chair — Kaohsiung Medical University; Ming-Ju Wu, Dr., Study Chair — Taichung Veterans General Hospital; Kuo-Cheng Lu, Dr., Principal Investigator — Taipei Buddhist Tzu Chi Medical Foundation; Lin-Kuo Ko, Dr., Study Chair — Taichung Tzu Chi Hospital; Jian-Lin Lu, Dr., Study Chair — Fu Jen Catholic University Hospital
Locations (7):
- Taiwan (7):
  - Kaohsiung Medical University Hospital, Kaohsiung City
  - Taipei Tzu Chi Hospital, New Taipei City
  - Fu Jen Catholic University Hospital, New Taipei City
  - Taichung Veterans General Hospital, Taichung
  - Tungs' Taichung MetroHarbor Hospital, Taichung
  - Tri-Service General Hospital, Taipei
  - Chang-Gung Memorial Hospital, Taoyuan District

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Simonsen E, Komenda P, Lerner B, Askin N, Bohm C, Shaw J, Tangri N, Rigatto C. Treatment of Uremic Pruritus: A Systematic Review. Am J Kidney Dis. 2017 Nov;70(5):638-655. doi: 10.1053/j.ajkd.2017.05.018. Epub 2017 Jul 15. PMID 28720208
- [Background] Malekmakan L, Tadayon T, Pakfetrat M, Mansourian A, Zareei N. Treatments of uremic pruritus: A systematic review. Dermatol Ther. 2018 Sep;31(5):e12683. doi: 10.1111/dth.12683. Epub 2018 Aug 23. PMID 30141218
- [Background] Niwa T, Emoto Y, Maeda K, Uehara Y, Yamada N, Shibata M. Oral sorbent suppresses accumulation of albumin-bound indoxyl sulphate in serum of haemodialysis patients. Nephrol Dial Transplant. 1991;6(2):105-9. doi: 10.1093/ndt/6.2.105. PMID 1906999
- [Background] Liu WC, Tomino Y, Lu KC. Impacts of Indoxyl Sulfate and p-Cresol Sulfate on Chronic Kidney Disease and Mitigating Effects of AST-120. Toxins (Basel). 2018 Sep 11;10(9):367. doi: 10.3390/toxins10090367. PMID 30208594
- [Result] Sukul N, Speyer E, Tu C, Bieber BA, Li Y, Lopes AA, Asahi K, Mariani L, Laville M, Rayner HC, Stengel B, Robinson BM, Pisoni RL; CKDopps and CKD-REIN investigators. Pruritus and Patient Reported Outcomes in Non-Dialysis CKD. Clin J Am Soc Nephrol. 2019 May 7;14(5):673-681. doi: 10.2215/CJN.09600818. Epub 2019 Apr 11. PMID 30975656